CLINICAL TRIAL: NCT03756753
Title: The RAPID Trial: Randomized Controlled Trial Assessing Point-of-care Influenza and Other Respiratory Virus Diagnostics
Brief Title: The RAPID Trial: Assessing Point-of-care Influenza and Other Respiratory Virus Diagnostics
Acronym: RAPID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Biofire (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 18-1492
Record Dates: First submitted 2018-11-27; First posted 2018-11-28 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Respiratory Pathogens; Upper Respiratory Tract Illness; Lower Respiratory Tract Illness; Acute Respiratory Infection

STUDY DESIGN:
Intervention Model Description: Participants will be allocated 1:1 by computer-generated randomization to either the intervention group - test result available to providers, or the control group- test result not available (routine clinical care).
Masking Description: Patients will be enrolled in the study, and will not initially know their study arm. After enrollment, the professional research assistant (PRA) will find out the study arm. Providers will be notified of the results for the intervention group. Providers are able to let patients know of their results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group- results known (Experimental): Providers of patients enrolled in this arm of the study will be notified of the point of care respiratory testing results
  Interventions: Diagnostic Test: Results available to provider
- Control group- results not known (No Intervention): Providers of patients enrolled in the study will not be notified of the point of care respiratory testing results

INTERVENTIONS:
Diagnostic Test: Results available to provider — Results of point of care testing are given to provider
  Arms: Intervention group- results known

SUMMARY:
The RAPID trial is a randomized controlled trial that looks at the clinical impact of a rapid respiratory test in a pediatric emergency department. Participants will be randomized to the intervention group - results available to medical providers, or the control group- results not available to medical providers.

DETAILED DESCRIPTION:
The RAPID trial is a randomized controlled trial of rapid respiratory viral testing in children presenting to an Emergency Department setting with acute respiratory symptoms. The patient cohort will be children 1 month to 18 years of age presenting to the Children's Hospital Colorado (CHCO) Emergency Department with influenza like illness who are triaged as level 3, 4, or 5 by the Emergency Severity Index, representing the typical patient population who are evaluated in an urgent care setting. All eligible participants will undergo a nasopharyngeal swab and point of care testing, and participants will be allocated 1:1 by computer-generated randomization to either the intervention group - test result available to providers, or the control group- test result not available (routine clinical care). The investigators will compare the clinical outcomes between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Age 1 month to < 18 years
2. For children aged 1 month to 12 months of age: Presentation to the study sites with temperature > 37.8°C or cough, sore throat, runny nose or nasal congestion
3. For children aged > 1 year to 18 years of age: Presentation to the study sites with influenza like illness, defined as temperature of >37.8⁰C and at least one of the following: cough, sore throat, runny nose or nasal congestion
4. Triage Level 3,4,5 based on Emergency Severity Index (refer to Appendix B for algorithm)

Exclusion Criteria:

1. Respiratory symptom duration > 14 days
2. Previous enrollment in study within past 14 days
3. Nurse-only visit
4. Triage levels 1 and 2 based on Emergency Severity Index

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 913 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of children prescribed an antibiotic at the Emergency Department (ED) visit | day 0
  Proportion of children who are prescribed an antibiotic at the ED visit.

SECONDARY OUTCOMES:
Proportion of children treated with influenza antiviral at the ED visit | day 0
  Proportion of patients treated with influenza antiviral at the ED visit in which a subject is enrolled in the study.
Proportion of patients who test positive for influenza treated with influenza antiviral at the ED visit | day 0
  Proportion of patients who test positive for influenza treated with influenza antiviral at the ED visit in which a subject is enrolled in the study.
ED length of stay (hours) | day 0
  Length of stay (in hours) in emergency department at the visit in which a subject is enrolled in the study.
Days of Hospitalization | day 0-10
  Proportion of patients hospitalized within 10 days of enrollment in the study
Number of repeat ED visits | day 0-10
  Number of repeat ED visits within 10 days of enrollment in the study
Number of tests ordered | day 0
  Number of tests ordered (labs, imaging, microbiologic testing) during visit in which a subject is enrolled in the study.
Relative clinical charges | day 0
  Relative clinical charges for ED visit in which a subject is enrolled in the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rao S, Lamb MM, Moss A, Mistry RD, Grice K, Ahmed W, Santos-Cantu D, Kitchen E, Patel C, Ferrari I, Dominguez SR. Effect of Rapid Respiratory Virus Testing on Antibiotic Prescribing Among Children Presenting to the Emergency Department With Acute Respiratory Illness: A Randomized Clinical Trial. JAMA Netw Open. 2021 Jun 1;4(6):e2111836. doi: 10.1001/jamanetworkopen.2021.11836. PMID 34086034